CLINICAL TRIAL: NCT01726621
Title: A User Evaluation of the MiniMed® 620G and 640G Insulin Pumps and Guardian® Link Transmitter
Brief Title: User Evaluation of the MiniMed 620G and 640G Insulin Pumps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CEP267
Record Dates: First submitted 2012-11-08; First posted 2012-11-15 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin dependent diabetics (Other): Subjects currently using an insulin pump transferred to use the Medtronic MiniMed 620G and 640G insulin pumps and Guardian Link transmitter
  Interventions: Device: Medtronic MiniMed 620G or 640G Insulin Pump

INTERVENTIONS:
Device: Medtronic MiniMed 620G or 640G Insulin Pump — Subjects to use the Medtronic MiniMed 620G or 640G Insulin Pump and Guardian Link transmitter to manage their diabetes for 4 - 6 weeks.

SUMMARY:
This six center international study will include two United Kingdom National Health Service centers, two centers in Melbourne, Australia and one center each in Denmark and Spain. The objective of the study is to evaluate subject acceptance of the a new insulin pump and transmitter together with the accompanying training materials. Descriptive data from participant questionnaires and device uploads will be evaluated.

Pediatric subjects between the ages of 7 - 18 years and adults from the age of 19 years of age upwards, who currently use an insulin pump in the management of their type 1 or type 2 diabetes, will be invited to participate. Each subject will be trained on the study device and then use it for approximately six weeks. During this time there will be three in-clinic visits and four follow-up phone calls, scheduled at the subjects' convenience. At the end of this period, they will revert back to their original insulin pump and complete a questionnaire on the study pump training materials, features and usability.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 7 years or older at time of screening
* Subject is current insulin pump user for at least 3 months
* Subject has the following Continuous Glucose Monitoring experience as determined by the Investigator:

  * Has experience and is able to insert/change sensor by herself/himself and
  * Has experience and can recharge the transmitter and
  * Has experience and can read sensor data in real-time on her/his pump screen
* Subject has signed a Patient Informed Consent form and is willing to comply with the study procedures;
* Subject is willing to complete study questionnaires throughout the study
* Must have one of the following clinical diagnosis:

  * Type 1 diabetes, for a minimum of 6 months prior to enrollment
  * Insulin requiring type 2 diabetes, for a minimum of 6 months prior to enrollment

Exclusion Criteria:

* Female subject has a positive urine pregnancy screening test.
* Female subject who plans to become pregnant during the course of study. If a woman becomes pregnant during participation, she will be withdrawn
* Subject has any condition that, in the opinion of the Investigator or qualified Investigational Center staff, may preclude him/her from participating in the study and completing study related procedures.
* Subject has impaired vision or hearing problems that could compromise the handling of the device as determined by Investigator or qualified Investigational Center staff
* Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks.

Ages: 7 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pratik Choudhary, MBBS, MRCP, Principal Investigator — King's College London
Locations (6):
- Australia (2):
  - St Vincent Hospital and The University of Melbourne, Fitzroy
  - The Royal Melbourne Hospital, Patkville
- Herlev Hospital, Herlev, Denmark
- Barcelona University Hospital, Barcelona, Spain
- United Kingdom (2):
  - University College Hospital, London
  - King's College London, London

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insulin Dependent Diabetics
Started | 55
Completed | 51
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Insulin Depedent Diabetics: Subject is current insulin pump user and has CGM experience as determined by the investigator.
Arm/Group | Insulin Depedent Diabetics
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 36
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (16.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: User Acceptance of the New MiniMed 620G and 640G Insulin Pumps and Guardian Link Transmitter
Description: Descriptive summary will be used to characterize the results of the study questionnaires. The questionnaire will use a Likert scale (rating of 1 to 7) to assess overall subject acceptance of the MiniMed 620G, 640G, and Guardian Link Transmitter. A response of 4 or greater on the Likert scale will be considered positive and indicate and product acceptance.
Time Frame: Four weeks of pump wear
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Insulin Depedent Diabetics
Number analyzed (Participants) | 55
units on a scale | 5.88 (1.32)

ADVERSE EVENTS:
Arm/Group | Insulin Dependent Diabetics
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 16/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Dependent Diabetics (N=55)
Bleeding cannula site (Skin and subcutaneous tissue disorders) | 1 (1)
Cough with sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Hyperglycaemia (Endocrine disorders) | 1 (1)
Insulin infusion set insertion site - bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Ketonemia (Endocrine disorders) | 1 (1)
Pyrexia (Immune system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Severe hypoglycemia (Endocrine disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation from Enlite sensor tape (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Urinary infection (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other